CLINICAL TRIAL: NCT00385892
Title: Feasibility Study DK150OS. Testing of Compression Textile. A Safety Study Among Healthy Volonteers
Brief Title: Safety Study of Textile Binder for Abdominal Compression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK150OS
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Healthy
Keywords: Healthy volonteers; Abdominal binder; IAP; MAP; APP

INTERVENTIONS:
Device: Abdominal binder

SUMMARY:
This safety study was carried out to investigate to what extent the use of an abdominal binder influences IAP. The study was designed as a comparative cross-over study measuring bladder pressure.

DETAILED DESCRIPTION:
Study Description: Transabdominal surgery might be associated with incisional pain, fear of rupture, inhibited mobilisation and risk of incisional herniation. An abdominal binder was developed for postoperative support of abdominal incisions. The abdominal binder provides a pressure of 10-15 mmHg.

Worlds Society on Abdominal Compartment Syndrome (WSACS) defines that Normal Intra-Abdominal Pressure (IAP) is approximately 5-7 mmHg in critically ill adults, and that Intra-Abdominal Hypertension (IAH) is a sustained or repeated pathologic elevation of IAP >12 mmHg. This safety study was carried out to investigate to what extent the use of the abdominal binder influences IAP. The study was designed as a comparative cross-over study measuring bladder pressure (Foley manometer, Holtec Medical, Copenhagen) in 11 healthy volunteers with and without wearing the abdominal binder.

Results IAP measurements without wearing the abdominal binder were found to be surprisingly high with a range between 8,0 and 16,7 mmHg. (mean 10,5 mmHg.). This finding is explained by the fact that the subjects were not under relaxation and the fact that half of the subjects according to their BMI were categorised as being overweight or fat. Other investigations have demonstrated that relaxation decreases IAP and that BMI is positively related to IAP.

We found that wearing the abdominal binder did increase IAP with a mean of 4,0 mmHg. (+/-1,4) or 39,3% (+/-14,61%).

In conclusion Relating our results to the WSACS guidelines regarding IAP and IAH it is not likely that the use of the abdominal binder will increase IAP to a clinically critical extent in patients with normal IAP. It must though be assessed from case to case, whether the use of the abdominal binder is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old
* Healthy
* Negative test of blood, nitrate or leucocytes in urinre
* Waist line measurement 97-110 cm

Exclusion Criteria:

* Pregnant
* Known allergy
* Know bladder disease
* Tendency of/clinicla symptoms of urinay infection
* Abdominal or urinary surgery
* Medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11
Dates: Start 2005-08; Study Completion 2005-10

PRIMARY OUTCOMES:
Intra Abdominal Pressure (IAP)
Mean Arterial Pressure (MAP)
Abdominal Perfussion Pressure (APP)

SECONDARY OUTCOMES:
Comfort
Freedom of movement

CONTACTS AND LOCATIONS:
Overall Officials: Lone M Poulsen, Consultant, Principal Investigator — ITA 303 KAS-Gentofte Niels Andersensvej 65 2900 Hellerup DENMARK